CLINICAL TRIAL: NCT07175207
Title: Study on the Safety and Efficacy of Umbilical Cord Blood Mononuclear Cells in the Treatment of Chronic Radiation Enteritis
Brief Title: Study on Safety and Efficacy of UCB-MNCs for Chronic Radiation Enteritis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Ji Zhu, Principal Investigator, Zhejiang Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025&UCB-MNCs&CRE
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Chronic Radiation Induced Intestinal Injury; Chronic Radiation Enteritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- UCB-MNCs (Experimental): UCB-MNCs are obtained from umbilical cord blood by density gradient centrifugation
  Interventions: Biological: UCB-MNCs

INTERVENTIONS:
Biological: UCB-MNCs — UCB-MNCs will be administered via intravenous infusion three times, once per week, with a dose of 3×10⁸ cells per infusion.

SUMMARY:
This study aims to evaluate the safety and efficacy of the umbilical cord blood mononuclear cells (UCB-MNCs) therapy for chronic radiation enteritis (CRE) by observing factors related to the therapeutic effect and adverse reactions of UCB-MNCs in treating CRE.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, with no restriction on gender;
2. History of pelvic and abdominal radiotherapy;
3. Patients diagnosed with chronic radiation-induced intestinal injury (CRII) via colonoscopy and pathological examination (≥3 months after the end of radiotherapy);
4. Diagnosed with grade 2-3 radiation-induced intestinal injury based on the clinical symptom assessment (RTOG classification) in Expert Consensus on Integrated Traditional Chinese and Western Medicine Diagnosis and Treatment of Radiation-Induced Intestinal Injury in China;
5. Poor response to conventional treatment for two weeks, with symptoms showing no remission or progressive aggravation;
6. Well-controlled tumor for ≥3 months;
7. No significant abnormalities in liver and renal function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the upper limit of normal (ULN); serum creatinine (Cr) and blood urea nitrogen (BUN) ≤ 2 times the upper limit of normal (ULN);
8. Expected lifespan of the subject ≥ 3 months;
9. The patient is informed of the study details and voluntarily signs the informed consent form;
10. Willing and able to receive treatment and complete follow-up in accordance with the protocol requirements, and able to adhere to the doctor's advice for basic treatment.

Exclusion Criteria:

1. Severe cardiac insufficiency (e.g., NYHA classification Grade Ⅲ or Ⅳ) and uncontrolled hypertension with medication (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 110 mmHg);
2. Positive results for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or syphilis;
3. Eastern Cooperative Oncology Group (ECOG) performance status score ≥ 2;
4. Currently participating in another clinical trial or having participated in another clinical trial within 4 weeks;
5. Patients with an allergic diathesis or known allergy to the preparation used in this trial;
6. Patients with comorbid mental illness who are unable to cooperate with treatment;
7. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Vienna Rectoscopy Score (VRS) | At 3 and 12 months after the last treatment.
  The VRS evaluates four core endoscopic features (mucosal hyperemia/erythema, mucosal ulceration, mucosal fibrosis/stenosis, and telangiectasia), with each feature scored on a 0-3 scale (0 = no abnormality, 3 = severe abnormality). The total VRS score is the sum of scores from the four features, typically ranging from 0 to 12. The total score directly reflects the severity of radiation-induced intestinal injury.

SECONDARY OUTCOMES:
Clinical remission rate | At 1 week, 1 month, 3 months, 6 months, and 12 months after the last treatment.
  Symptoms such as hematochezia and diarrhea will be counted before treatment and at 1 week, 1 month, 3 months, 6 months, and 12 months after the last treatment. The corresponding symptom remission rate will be calculated by comparing with the pre-treatment status.
Change from baseline LENT-SOMA scoring scale | At 3 months and 12 months after the last treatment.
  LENT-SOMA uses a 0-4 grading system for each of the four dimensions (subjective, objective, management, analytic), with scores directly reflecting the severity of radiation-induced tissue injury. A higher LENT-SOMA grade indicates more severe radiation-induced tissue damage.
Change from baseline visual analog scale (VAS) | At 1 week, 1 month, 3 months, 6 months, and 12 months after the last treatment.
  VAS is a simple tool to measure pain extent: it uses a 10-centimeter horizontal line, with "no pain at all" marked at 0 and "worst pain imaginable" at 10. Patients mark a point matching their current pain.
Hemoglobin concentration | Changes in hemoglobin levels will be compared before treatment and at 1 week, 1 month, 3 months, 6 months, and 12 months after the last treatment.
Changes in Intestinal Flora Distribution | At 1 week and 1 month after the last treatment.
  Intestinal flora distribution specifically describes the composition, quantity, and proportional balance of the microbial species.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No